CLINICAL TRIAL: NCT01727609
Title: A Multi-centre Randomised Controlled Trial of Two Speeds of Daily Increment of Milk Feeding in Very Preterm or Very Low Birth Weight Infants
Brief Title: Speed of Increasing Milk Feeds Trial
Acronym: SIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIFT01
Record Dates: First submitted 2012-10-11; First posted 2012-11-16 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2018-07

CONDITIONS: Premature Birth; Late-onset Invasive Infection; Necrotizing Enterocolitis
Keywords: Preterm; Very low birth weight; Feeding; Enteral; Milk; Sepsis; Necrotizing enterocolitis (NEC)
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing; Sepsis | interventions — Milk, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Slower milk feed increment (Active Comparator): Increase milk feeds by 18 ml/kg/day until on full milk feeds (tolerating 150 ml/kg/day for 3 consecutive days)
  Interventions: Dietary Supplement: Milk feed (breast milk or formula milk)
- Faster milk feed increment (Experimental): Increase milk feeds by 30 ml/kg/day until on full milk feeds (tolerating 150 ml/kg/day for 3 consecutive days)
  Interventions: Dietary Supplement: Milk feed (breast milk or formula milk)

INTERVENTIONS:
Dietary Supplement: Milk feed (breast milk or formula milk)

SUMMARY:
Survival of preterm infants has increased greatly over the years, so a major aim now is to improve the long term outlook for these babies and to avoid serious complications. The way babies are fed in early life affects short and long-term health and survival.

Because the bowels of preterm infants have not matured, they cannot digest large volumes of milk feeds straight away. Until the gut matures, nutrition is provided by intravenous drip while the amount of milk given is gradually increased over time. Increasing the amount of milk rapidly may increase the risk of gut complications. Increasing the amount of milk given more slowly means that intravenous nutrition is needed for longer; there is an associated risk of infection proportional to the time the intravenous line is present in the bloodstream of these infants. Despite the importance of milk feeding preterm infants, there have been few studies to inform how best to balance these risks, and what the best way to increase feeds in these infants is - this study sets out to address this missing information.

The study will compare two different speeds of milk feed increase, one 'faster' and one 'slower', both within rates currently used in United Kingdom neonatal units. The study aims to find out if either speed of milk feed increase gives better outcomes for the infants. Investigators will measure a variety of outcomes, such as survival without disability, infection, bowel problems, growth and long-term physical and mental development, as well as the impact on families and the National Health Service, including costs.

The study is being led by an established team of researchers who have run similar studies before, and uses an established network of neonatal units that have taken part in previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth <32 weeks, or birth weight less than 1,500 g
* Receiving ≤30 ml/kg/day of milk at randomisation
* Written informed parental consent is obtained

To ensure the widest applicability to preterm infants across the United Kingdom, those exclusively breast milk fed, formula milk fed, or receiving mixed feeds will be included

Exclusion Criteria:

* Infants with a severe congenital anomaly
* Infants who, in the opinion of the treating clinician, have no realistic chance of survival
* Infants who are unlikely to be traceable for follow-up at 24 months of age corrected for prematurity (for example, infants of non-United Kingdom residents)

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2804 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Survival without moderate or severe disability | 24 months of age corrected for prematurity

SECONDARY OUTCOMES:
Survival to discharge home | Participants will be followed from trial entry until hospital discharge (typically at 36 corrected weeks' gestation), an expected average of 8 weeks.
Incidence of microbiologically-confirmed or clinically suspected late-onset invasive infection | Participants will be followed from trial entry until hospital discharge (typically at 36 corrected weeks' gestation), an expected average of 8 weeks.
Incidence of necrotizing enterocolitis (Bell stage 2 or 3) | Participants will be followed from trial entry until hospital discharge (typically at 36 corrected weeks' gestation), an expected average of 8 weeks.
Time taken to reach full milk feeds (tolerating 150 ml/kg/day for 3 consecutive days) | Participants will be followed from trial entry until hospital discharge (typically at 36 corrected weeks' gestation), an expected average of 8 weeks.
Growth (weight and head circumference) at hospital discharge | Participants will be followed from trial entry until hospital discharge (typically at 36 corrected weeks' gestation), an expected average of 8 weeks.
  Measured by weight and head circumference z-scores
Duration of parenteral feeding before hospital discharge | Participants will be followed from trial entry until hospital discharge (typically at 36 corrected weeks' gestation), an expected average of 8 weeks.
Length of time in intensive care | Participants will be followed from trial entry until hospital discharge (typically at 36 corrected weeks' gestation), an expected average of 8 weeks.
Length of hospital stay | Participants will be followed from trial entry until hospital discharge (typically at 36 corrected weeks' gestation), an expected average of 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Dorling, MBChB DCH MD, Principal Investigator — Division of Neonatal-Perinatal Medicine, Dalhousie University, Halifax, NS, Canada
Locations (57):
- National Maternity Hospital, Dublin, Dublin, Ireland
- United Kingdom (56):
  - William Harvey Hospital, Ashford
  - Royal Maternity Hospital, Belfast, Belfast
  - Birmingham Women's Hospital, Birmingham
  - Birmingham City Hospital, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Southmead Hospital, Bristol
  - St Michael's Hospital, Bristol
  - St Peters Hospital, Chertsey
  - Countess of Chester Hospital, Chester
  - University Hospital Coventry, Coventry
  - Leighton Hospital, Crewe
  - Derbyshire Children's Hospital, Derby
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Princess Royal Maternity Hospital, Glasgow, Glasgow
  - Southern General Hospital, Glasgow
  - Gloucestershire Royal Hosptial, Gloucester
  - Calderdale Royal Hospital, Halifax
  - Hull Royal Infirmary, Hull
  - Kettering General Hospital, Kettering
  - Leeds General Infirmary, Leeds
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Lincoln County Hospital, Lincoln
  - St George's Hospital, London
  - Altnagelvin Area Hospital, Londonderry
  - James Cook University Hospital, Middlesbrough
  - Royal Victoria Infirmary, Newcastle
  - Northampton General Hospital, Northampton
  - Nottingham City Hospital, Nottingham
  - Queen's Medical Centre, Nottingham
  - John Radcliffe Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Craigavon Area Hospital, Portadown
  - Queen Alexandra Hospital, Portsmouth, Portsmouth
  - Royal Berkshire Hospital, Reading
  - Queen's Hospital, Romford, Romford
  - Jessop Wing, Sheffield, Sheffield
  - Royal Shrewsbury Hospital, Shrewsbury
  - Princess Anne Hospital, Southampton, Southampton
  - University Hospital of North Tees, Stockton-on-Tees
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Sunderland Royal Hospital, Sunderland
  - King's Mill Hospital, Sutton in Ashfield
  - Singleton Hospital, Swansea
  - Great Western Hospital, Swindon, Swindon
  - Croydon University Hospital, Thornton Heath
  - Royal Cornwall Hospital, Truro
  - Arrowe Park Hospital, Wirral, Upton
  - Pinderfields General Hospital, Wakefield
  - Warrington Hospital, Warrington
  - Wishaw General Hospital, Wishaw
  - New Cross Hospital, Wolverhampton
  - Worcestershire Royal Hospital, Worcester
  - York Hospital, York